CLINICAL TRIAL: NCT07229027
Title: Global Overweight and oBesE (GLOBE) Patient Registry, Development and Implementation of Disease-specific: Severity, Quality of Life and Cost Instruments.
Acronym: GLOBE
Status: Recruiting | Type: Observational
Sponsor: Medialis Ltd. (Industry)
Responsible Party: Principal Investigator, Ravi Jandhyala, Dr, Medialis Ltd.
Other Study IDs: MED 63
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Overweight (BMI > 25); Obesity & Overweight
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We are conducting this study to develop a disease-specific instrument, a quality of life instrument and a comprehensive list of costs associated with overweight and obesity.

DETAILED DESCRIPTION:
Despite evidence on the burden of BMI >25, few disease-specific instruments comprehensively capture its multidimensional impact. Existing frameworks often target obesity (BMI ≥30) or patients on pharmacological or surgical therapy. Overweight and extremely obese populations are underrepresented, and economic and psychosocial dimensions are rarely integrated into severity staging.

This study, therefore, aims to systematically evaluate symptoms, comorbidities, HRQoL, and costs across the full spectrum of individuals with BMI >25, excluding those on GLP-1 therapy. Integrating clinician and patient perspectives will support the development of more inclusive severity measures and inform early intervention strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patient group

  1. Patient is aged ≥18 years at the time of survey completion.
  2. Patient has a BMI over 25 (self-reported)
  3. Patient is willing to participate in all study activities.
  4. Patient is able to read, write, and converse in English.
* Healthcare professional participant must meet the following criteria for inclusion in the study:

  1. HCP is aged ≥18 years at the time of survey completion.
  2. HCP is suitably qualified and involved in the healthcare management of patients with a BMI over 25
  3. HCP is willing to participate in all study activities.
  4. HCP is able to read, write, and converse in English.

     Exclusion Criteria:

A participant who meets any of the following criteria will be excluded from the study:

1. Participants do not have the cognitive capacity to provide informed consent.
2. Participants with severe co-morbidity that might affect study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with BMI over 25 Healthcare professionals treating patients.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Development of a Disease-Specific Questionnaire | 2 months

SECONDARY OUTCOMES:
Quality of Life Instrument | 2 months

OTHER OUTCOMES:
Cost Implications of Obesity | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Online recruitment, Milton Keynes, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT07229027/Prot_SAP_000.pdf